CLINICAL TRIAL: NCT07062939
Title: Comparative Effects of Manual Versus Mechanical Airway Clearance Techniques in Cystic Fibrosis
Brief Title: Comparative Effects of Mechanical and Manual Airway Clearance Techniques in Cystic Fibrosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0350
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Cystic Fibrosis
Keywords: postural drainage; flutter; pulmonary rehabilitation
MeSH Terms: conditions — Cystic Fibrosis | interventions — Drainage, Postural

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postural drainage with ACBT (Experimental): postural drainage and active cycle breathing technique for 2 times a day for 30 min for 4 weeks
  Interventions: Other: postural drainage with ACBT
- flutter with ACBT (Active Comparator): active cycle breathing technique with flutter for 30 min for 4 week and 2 times a day
  Interventions: Other: flutter with ACBT

INTERVENTIONS:
Other: postural drainage with ACBT — postural drainage and ACBT for 2 times a day for 30 min for 4 weeks.
  Arms: postural drainage with ACBT
Other: flutter with ACBT — flutter with active cycle breathing technique for 30 min. for 4 week and 2 times a day.
  Arms: flutter with ACBT

SUMMARY:
This study will help to establish evidence-based physiotherapy on postural drainage and ACBT against flutter with ACBT is better to improve sleep quality, adherence, dyspnea in patients with cystic fibrosis and which method can improve respiratory function, reduce the risk of complications after illness and additionally advancements in respiratory therapy can lead to improve sleep quality, individual preference and adherence and dyspnea.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a genetic disorder that leads to the accumulation of thick mucus in the lungs and other organs, resulting in recurrent infections and progressive lung damage. This condition is due to mutations in the cystic fibrosis transmembrane conductance regulator CFTR gene, which governs the transport of chloride and other ions across cell membranes. CF affects a significant number of people worldwide, with certain genetic mutations leading to more severe manifestations of the disease. The management of CF is centered on clearing the airways of mucus to prevent infections and slow the progression of lung damage. Various studies have yielded inconsistent results regarding the comparative effectiveness of manual versus mechanical airway clearance techniques in improving pulmonary function tests (PFTs) in CF patients.

Despite the existing literature on postural drainage with ACBT in patient with cystic fibrosis, there is a significant research gap regarding the flutter and ACBT on the bases of outcomes in cystic fibrosis. Most studies have not adequately addressed the distinct needs and responses of flutter with ACBT on the basis of outcomes, leaving a void in understanding how these two intervention effect on sleep, adherence and dyspnea in the context of patients with cystic fibrosis. Closing this gap is essential for developing evidence-based and pulmonary rehabilitation techniques for this specific patient group.

ELIGIBILITY:
Inclusion Criteria:

* Patient having clinically diagnose Cystic fibrosis.
* Age 16-40 year.
* Both male and female.
* Subjects who are conscious and cooperative .

Exclusion Criteria:

* Rib fracture
* History of cardiac surgery.
* Subject with any Physical or Mental Disability
* Age less than 16 years

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-07-06 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 4 weeks
  This is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval, show the sleep quality duration and efficacy. Many of the aforementioned research employed the PSQI, the most commonly utilized sleep quality index. the validity and reliability of the PSQI in healthcare professionals, or even in high-pressure shift employees. The PSQI's validity and reliability in regularly planned, low-pressure groups, such as adults in good health who live in the vicinity, differed greatly from front-line COVID-19 healthcare personnel. The conventional test theory (CTT) serves as the primary foundation for the reliability and validity research on PSQI. While there is little to no link between the PSQI and problems including anger, nausea,stiffness, and urinary disorder, it does have a strong correlation with the Insomnia Severity Index, polysomnography, and other sleep quality indicators
The Shwachman-Kulczycki score | 4 weeks
  This is the first scoring system used in cystic fibrosis to assess disease severity and show the adherence to treatment. In the present study, the total Shwachman-Kulczycki score correlated positively with the scores for each of its four domains, and physical activity was the aspect that most influenced total score.
Borg dyspnea scale | 4 weeks
  The instruments provide a standard method for patients to select ratings of dyspnea on a scale based on descriptors that correspond to specific numbers

SECONDARY OUTCOMES:
The Breathlessness, Cough and Sputum Scale (BCSS) | 4 weeks
  This scale is used to predict patient exacerbations by evaluating common symptoms, Results suggest BCSS scores are valid indicators of the severity of cough and sputum in patients with COPD. Scores for both items were correlated with sputum volume.

CONTACTS AND LOCATIONS:
Overall Officials: iram nawaz, mphill, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital, Sheikhupura, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zisi D, Chryssanthopoulos C, Nanas S, Philippou A. The effectiveness of the active cycle of breathing technique in patients with chronic respiratory diseases: A systematic review. Heart Lung. 2022 May-Jun;53:89-98. doi: 10.1016/j.hrtlng.2022.02.006. Epub 2022 Feb 27. PMID 35235877
- [Background] Chen Q, Shen Y, Zheng J. A review of cystic fibrosis: Basic and clinical aspects. Animal Model Exp Med. 2021 Sep 16;4(3):220-232. doi: 10.1002/ame2.12180. eCollection 2021 Sep. PMID 34557648
- [Background] Elborn JS, Ramsey BW, Boyle MP, Konstan MW, Huang X, Marigowda G, Waltz D, Wainwright CE; VX-809 TRAFFIC and TRANSPORT study groups. Efficacy and safety of lumacaftor/ivacaftor combination therapy in patients with cystic fibrosis homozygous for Phe508del CFTR by pulmonary function subgroup: a pooled analysis. Lancet Respir Med. 2016 Aug;4(8):617-626. doi: 10.1016/S2213-2600(16)30121-7. Epub 2016 Jun 10. PMID 27298017
- [Background] Wilson LM, Saldanha IJ, Robinson KA. Active cycle of breathing technique for cystic fibrosis. Cochrane Database Syst Rev. 2023 Feb 2;2(2):CD007862. doi: 10.1002/14651858.CD007862.pub5. PMID 36727723
- [Background] Rowbotham NJ, Smith SJ, Davies G, Daniels T, Elliott ZC, Gathercole K, Rayner OC, Smyth AR. Can exercise replace airway clearance techniques in cystic fibrosis? A survey of patients and healthcare professionals. J Cyst Fibros. 2020 Jul;19(4):e19-e24. doi: 10.1016/j.jcf.2019.10.026. Epub 2019 Nov 15. PMID 31740105
- [Background] Zhao M, Cheng L, Fu W, Ma X, Chen X. Measuring parents' perceptions of inclusive school quality in China: the development of the PISQ scale. Int J Dev Disabil. 2021 Mar 10;68(6):824-837. doi: 10.1080/20473869.2021.1895696. eCollection 2022. PMID 36568612